CLINICAL TRIAL: NCT05177913
Title: Assessment of Factors Influencing Parents' Attendance Time During Feeding Time of Premature Infants Born Before 35 Weeks of Amenorrhea in Besançon University Hospital
Acronym: PréPaLim
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: P/2019/409
Record Dates: First submitted 2021-09-14; First posted 2022-01-05 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Premature Birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The precise description of parental presence and the associated factors will make it possible to construct an intervention in order to correct potentially low parental participation. The demonstration of the effectiveness of such an intervention will be the subject of a larger study (PHRIP type). Ultimately, the investigators want to personalize the daily support for parents to offer optimal support for parenting.

DETAILED DESCRIPTION:
Considering the importance of the bond of attachment, and in particular the emotional tuning between the adult and the premature baby and the particularly important interactions during feeding, it seemed essential to us to make an evaluation of the parental presence during the meals. , which sheds light on the factors influencing this presence.

The presence time seems to vary depending on: the child's background, the profile of the parents, the profile of the child and environmental factors.

Knowing the factors influencing this presence is essential in order to understand the obstacles to the arrival of parents, to think as a team and to offer personalized support in order to allow them to be more present with their baby.

ELIGIBILITY:
Inclusion Criteria:

* Premature newborn under 35 weeks of amenorrhea (AS), hospitalized at Besançon University Hospital,
* Newborn baby whose parents:

expressed their non-opposition to participate in the study, are affiliated to a social security scheme, are of age, express themselves easily in French.

Exclusion Criteria:

* Newborn baby whose parents object to participating in the study,
* Newborns presenting severe malformative anomalies, or malformations of the oral sphere,
* Newborn baby whose transfer is scheduled before the end of hospitalization (excluding birthing pool at the CHU de Besançon).

Ages: 1 Day to 10 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The premature newborn born before 35 weeks of amenorrhea at the Besançon University Hospital and his parents (birth couple).
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2021-09-16 (Actual); Primary Completion 2023-05-26 (Actual); Study Completion 2023-05-26 (Actual)

PRIMARY OUTCOMES:
The time of parental presence | Up to 6 months
  Quantify the time of parental presence during the meals of premature children born before 35 weeks of amenorrhea (AS)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Besancon, Besançon, France